CLINICAL TRIAL: NCT00199082
Title: Multicenter Study to Optimise Therapy of B-ALL, Burkitt's NHL and High-Grade Non-Hodgkin's Lymphoma in Adults (Amend 7)
Brief Title: Newly Diagnosed Mature B-ALL, Burkitt's Lymphoma and Other High-grade Lymphoma in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nicola Goekbuget (Other)
Responsible Party: Sponsor-Investigator, Nicola Goekbuget, Study Coordinator, Goethe University
Organization: Goethe University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL05
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Burkitt's Lymphoma; Burkitt's Leukemia; Mediastinal Neoplasms; Lymphoblastic Lymphoma; Large Cell Anaplastic Lymphoma
Keywords: High-grade NHL; De novo; Mature B-ALL; Burkitt'S NHL; Chemotherapy; Rituximab; Primary mediastinal diffuse large cell lymphoma; B-precursor lymphoblastic lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Mediastinal Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Doxorubicin; Cyclophosphamide; Cytarabine; Dexamethasone; Prednisolone; Etoposide; Ifosfamide; Methotrexate; Granulocyte Colony-Stimulating Factor; Rituximab; Vincristine; Vindesine; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): This is a single arm trial with complex chemotherapy (6 cycles) stratified by age, subtype (Burkitt-leukemia vs Burkitt-lymphoma) and initial involvement
  Interventions: Drug: Adriamycin; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone/Prednisolone; Drug: VP16; Drug: Ifosfamide; Drug: Methotrexate; Drug: G-CSF; Drug: Rituximab; Drug: Vincristine/Vindesine; Procedure: Irradiation (in specific conditions)

INTERVENTIONS:
Drug: Adriamycin
Drug: Cyclophosphamide
Drug: Cytarabine
Drug: Dexamethasone/Prednisolone
Drug: VP16
Drug: Ifosfamide
Drug: Methotrexate
Drug: G-CSF
Drug: Rituximab
Drug: Vincristine/Vindesine
Procedure: Irradiation (in specific conditions)

SUMMARY:
The study evaluates the efficacy and tolerability of alternating short cycles of high-dose and conventional chemotherapy in combination with rituximab in CD20 positive patients, followed by local radiation therapy in the case of initial mediastinal or central nervous system (CNS) involvement or a residual tumor after chemotherapy. A dose-reduced regimen is offered for patients estimated to be over 55 years, biologically.

ELIGIBILITY:
Inclusion Criteria:

* Burkitt's leukemia or Burkitt's lymphoma or primary mediastinal large B-cell lymphoma or B-precursor lymphoblastic lymphoma or large cell anaplastic lymphoma
* Age > 15 years
* Written informed consent

Exclusion Criteria:

* Serious secondary diseases, including psychiatric conditions, under which the required therapy compliance is not to be expected
* HIV infection
* Secondary lymphoma following prior chemotherapy/radiotherapy or active second malignancy
* Known severe allergy to foreign proteins
* Pre-treatment other than 1 cycle CHOP or similar; < 1 week of another chemotherapy.
* Pregnancy or nursing
* Participation in other studies that interfere with study therapy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2002-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Remission rate
Remission duration
Disease free survival
Overall survival

SECONDARY OUTCOMES:
Dose and time compliance
Toxicity according to National Cancer Institute (NCI)-Common Toxicity Criteria (CTC)
Death under therapy and in complete remission (CR)
Localisations of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Goekbuget, Dr. med., Principal Investigator — University Hospital of Frankfurt (Main)
Locations (1):
- University Hospital, Medical Dept. II, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoelzer D, Walewski J, Dohner H, Viardot A, Hiddemann W, Spiekermann K, Serve H, Duhrsen U, Huttmann A, Thiel E, Dengler J, Kneba M, Schaich M, Schmidt-Wolf IG, Beck J, Hertenstein B, Reichle A, Domanska-Czyz K, Fietkau R, Horst HA, Rieder H, Schwartz S, Burmeister T, Gokbuget N; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Improved outcome of adult Burkitt lymphoma/leukemia with rituximab and chemotherapy: report of a large prospective multicenter trial. Blood. 2014 Dec 18;124(26):3870-9. doi: 10.1182/blood-2014-03-563627. Epub 2014 Oct 30. PMID 25359988